CLINICAL TRIAL: NCT06423820
Title: Preoperative Ondansetron Lozenge for Prevention of Postoperative Nausea and Vomiting in Pediatrics Undergoing Squint Surgeries: A Randomized Controlled Trial
Brief Title: Preoperative Ondansetron Lozenge for Prevention of Postoperative Nausea and Vomiting in Pediatrics Undergoing Squint Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 36264PR640/4/24
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Ondansetron Lozenge; Postoperative Nausea and Vomiting; Pediatrics; Squint
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Strabismus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (Ondansetron lozenge) (Experimental): Pediatric patients will receive ondansetron lozenge 4 mg (Ondalenz ©), 2 hours before surgery as a study group.
  Interventions: Drug: Ondansetron lozenge
- Group C (Control) (No Intervention): Pediatric patients will not receive ondansetron as a control group.

INTERVENTIONS:
Drug: Ondansetron lozenge — Pediatric patients will receive ondansetron lozenge 4 mg (Ondalenz ©), 2 hours before surgery.
  Arms: Group S (Ondansetron lozenge)

SUMMARY:
The aim of this study is to evaluate the role of ondansetron lozenge on prevention of postoperative nausea and vomiting (PONV) in pediatrics undergoing squint surgeries.

DETAILED DESCRIPTION:
Post-operative nausea and vomiting (PONV) are two of the most common and distressing complications related to surgery and anesthesia.

In several studies PONV occurred in 13% to 42% of pediatric surgical patients, while severe cases are less common, occurring in 1-3% of patients. Volatile anesthetics are the main cause in the early post-operative period (0-2 h), with dose-response relationship. In the delayed post-operative period (2-24 h) the main predictors are childhood, PONV in the early period, and the use of postoperative opioids.

Ondansetron is generally considered to be the first-line antiemetic for patients because of its favorable side effect profile. Ondansetron reduces the activity of the vagus nerve, which deactivates the vomiting center in the medulla oblongata, and also blocks serotonin receptors in the chemoreceptor trigger zone, Ondansetron is an effective drug in the prevention and treatment of PONV by having low side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age from 4 to 15 years.
* American Society of Anesthesiology (ASA) physical status I, II.
* Pediatric patients undergoing squint surgeries.

Exclusion Criteria:

* Patients who had received any medication with antiemetic properties within 24 h before surgery.
* Post-operative period (for reasons other than rescue antiemetic therapy).
* Patients with known liver or renal disease.
* Patients with a history of vomiting or retching within 24 h before surgery.

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting | 24 hours postoperatively
  The incidence of postoperative nausea and vomiting (PONV) will be measured in the first 24 postoperative hours at the intervals of 0-2h (early PONV), 2-12h (delayed PONV), and 12- 24h (late PONV)

SECONDARY OUTCOMES:
Severity of postoperative nausea and vomiting (PONV) | 24 hours postoperatively
  The severity of postoperative nausea and vomiting (PONV) will be scored as follows: [0 = no nausea and no retching; 1 complaining of sickness and retching; vomiting one or two times in 30 min; and 3 vomiting more than two times in 30 min] in the first 24 hours postoperatively.
Number of emetic episodes | 24 hours postoperatively
  Number of emetic episodes will be measured from the end of surgery till 24 hours postoperatively.
Time to onset of emesis | 24 hours postoperatively
  Time to onset of emesis will be measured from the end of surgery till 24 hours postoperatively.
Incidence of oculo-cardiac reflex (OCR) | 24 hours postoperatively
  Incidence of oculo-cardiac reflex (OCR) will be recorded. OCR is defined as a 10-20% decrease in the resting heart rate and/or the occurrence of any arrhythmia.
Parental satisfaction | 24 hours postoperatively
  Degree of parental satisfaction by using an 11-pointverbal numeric scoring system (0 = not at all satisfied, 10 = fully satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.